CLINICAL TRIAL: NCT05389566
Title: Diabetes, Falls, and Fractures
Acronym: DIAFALL
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Nicklas Højgaard-hessellund Rasmussen, Postdoc and researcher, Aalborg University Hospital
Other Study IDs: N-20190004
Record Dates: First submitted 2022-05-06; First posted 2022-05-25 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Peripheral Neuropathy; Diabetes; Balance; Distorted; Vestibular Neuropathy; Muscle Weakness; Sarcopenia; Autonomic Neuropathy, Diabetic; Small Fiber Neuropathy
Keywords: Diabetes; Balance; Vestibular; Neuropathy; Muscle Weakness; Autonomic Neuropathy; Small Fiber Neuropathy; Postural control
MeSH Terms: conditions — Diabetes Mellitus; Vestibular Neuronitis; Muscle Weakness; Sarcopenia; Diabetic Neuropathies; Small Fiber Neuropathy | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type 1 diabetes: People with type 1 diabetes above 40 years
  Interventions: Diagnostic Test: Quantative Sensory Testing; Diagnostic Test: NCStat-DPN-Check; Diagnostic Test: Composite Autonomic Symptom Score 31; Diagnostic Test: Computerized dynamic posturography; Diagnostic Test: Video Head Impulse Test; Diagnostic Test: Accelerometer; Diagnostic Test: Handgrip strength; Diagnostic Test: Dual Energy X-ray Absorbtimetry scan; Diagnostic Test: Force Plate Platform
- People with type 2 diabetes: People with type 2 diabetes above 50 years
  Interventions: Diagnostic Test: Quantative Sensory Testing; Diagnostic Test: NCStat-DPN-Check; Diagnostic Test: Composite Autonomic Symptom Score 31; Diagnostic Test: Computerized dynamic posturography; Diagnostic Test: Video Head Impulse Test; Diagnostic Test: Accelerometer; Diagnostic Test: Handgrip strength; Diagnostic Test: Dual Energy X-ray Absorbtimetry scan; Diagnostic Test: Force Plate Platform
- Healthy controls: Healthy controls without diabetes
  Interventions: Diagnostic Test: Quantative Sensory Testing; Diagnostic Test: NCStat-DPN-Check; Diagnostic Test: Composite Autonomic Symptom Score 31; Diagnostic Test: Computerized dynamic posturography; Diagnostic Test: Video Head Impulse Test; Diagnostic Test: Accelerometer; Diagnostic Test: Handgrip strength; Diagnostic Test: Dual Energy X-ray Absorbtimetry scan; Diagnostic Test: Force Plate Platform

INTERVENTIONS:
Diagnostic Test: Quantative Sensory Testing — Evaluation of small fiber neuropathy
Diagnostic Test: NCStat-DPN-Check — Evaluation of large fiber neuropathy
Diagnostic Test: Composite Autonomic Symptom Score 31 — Evaluation of autonomic neuropathy
Diagnostic Test: Computerized dynamic posturography — Evaluation of dynamic postural control
  Other Names: Bertec
Diagnostic Test: Video Head Impulse Test — Evaluation of vertigo and the vestibular organ
  Other Names: V-Hit
Diagnostic Test: Accelerometer — Evaluation of gait pattern
  Other Names: Sens Innovation, Copenhagen Denmark
Diagnostic Test: Handgrip strength — Evaluation of muscle strength
  Other Names: Hydraulic dynamometer, Saehan Coorporation, Gyungnam, South Korea
Diagnostic Test: Dual Energy X-ray Absorbtimetry scan — Evaluation of body composition
  Other Names: Dexa, Hollogic Horizon (4500 Hollogic Inc., Marlborough, MA, USA)
Diagnostic Test: Force Plate Platform — Evaluation of balance while standing still
  Other Names: Plux Biosignals, S.A, Arruda dos Vinhos, Portugal

SUMMARY:
Comparing severity of diabetic peripheral neuropathy (small and large fibers including autonomic neuroapthy) to postural control and vestibular measurements

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with minimum 40 years of age and maximum 70 years of age.
2. Diagnosis of T1D or T2D
3. Diagnosis of diabetes with at least one year prior to inclusion of the study
4. Signed the informed consent.

Exclusion Criteria:

1. Severe decreased liver function (Alanin amino-transaminase (ALAT)>250u/l, GammaGlutamyltransferase (GGT)>150u/l)
2. Moderate to severe kidney dysfunction, estimated Glomerular Filtration Rate (eGFR) <15mmol/L/1,73m2
3. Pregnancy or breast feeding
4. Active malignancy or terminal ill.
5. Current or previous alcohol- or drug abuse

8. Not being able to understand Danish written and/or verbally 9. Terms according to investigators judgement that makes subjects unsuitable to participate including lack of understanding or reduced physical ability. 10. Participating in other clinical studies 11. Maximum of 10 hours of weekly exercise.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with type 1 or 2 diabetes from general practice or outpatient clinic at Steno Diabetes Center North Denmark
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Co-existence of peripheral- and vestiubular neuropathy in people with diabetes | through study completion, an average of 2 years
  Vestibular neuropathy (measured by pathological video head impulse test (v-Hit) (one-sided, two-sided or specific arcways)) will be compared with peripheral neuropathy (measured by quantitative sensory testing, nerve conduction and COMPASS-33) in the population with diabetes.
Co-existence of peripheral neuropathy and impaired dynamic postural control in people with diabetes | through study completion, an average of 2 years
  Dynamic balance (measured by Bertec) will be compared with peripheral neuropathy (measured by quantitative sensory testing, nerve conduction and COMPASS-33) in the population with diabetes.

SECONDARY OUTCOMES:
Correlation between the severity of peripheral neuropathy and the severity of vestibular in terms of degree of pathological video head impulse testingneuropathy | through study completion, an average of 2 years
  QST / NC-Stat DPNCheck vs v-Hit
Correlation between distal neuropathy and dynamic postural control (including patterns) | through study completion, an average of 2 years
  QST / NC-Stat DPNCheck vs accelerometer / Bertec
The impact of peripheral neuropathy on postural control (In quite stance) | through study completion, an average of 2 years
  QST / Correlation between muscle strength and peripheral neuropathy vs Force Plate

OTHER OUTCOMES:
Exploratory | through study completion, an average of 2 years
  accelerometer (SENS Innovation, Copenhagen, Denmark) measures (postural control during walking)
Exploratory | through study completion, an average of 2 years
  Correlations between different outcomes of Bertec and v-Hit vs peripheral neuropathy (all individual examinations and arcways)
Muscle strength and peripheral neuropathy | through study completion, an average of 2 years
  Correlation between muscle strength and peripheral neuropathy (DEXA-scans, hand grup strength, QST, Correlation between muscle strength and peripheral neuropathy

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Possible requirement for external data analysis

REFERENCES:
- [Derived] Mahalingasivam AA, Jespersen AK, Ejskjaer N, Hougaard DD, Vestergaard P, Rasmussen NH, Roikjer J. The co-existence of peripheral and vestibular neuropathy in diabetes: a cross-sectional study. Eur Arch Otorhinolaryngol. 2024 Feb;281(2):663-672. doi: 10.1007/s00405-023-08130-6. Epub 2023 Jul 29. PMID 37515636